CLINICAL TRIAL: NCT06021548
Title: Biopsychosocial Markers of Addiction in Opioid Users: an Integrated Approach
Acronym: BEBOP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8668
Record Dates: First submitted 2023-08-10; First posted 2023-09-01 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Opioid Use Disorder
Keywords: Psychiatry, Neurobiology, Epidemiology, Bioinformatics
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples will be taken by finger prick and blood collection (between 200 and 500 microliters per sample) on a capillary tube in order to avoid generating a craving by using phlebotomy to collect venous blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample — Finger stick blood spots will be collected at V0 and M12
Other: Saliva sample — Saliva sample will be collected at V0
Other: Hair sample — Hair sample will be collected at V0 (optional)

SUMMARY:
Opioid use disorder (OUD) is a chronic and severe psychiatric condition, defined by problematic opioid use, that significantly impairs interpersonal and social functioning. Over the last 10 years, a dramatic increase in the prevalence of OUD and deaths by overdose has occurred in several developed countries, in particular the USA. In France, similarly, the burden associated with OUD is worsening, and now represents a major public health crisis. During last decades, it has been demonstrated that OUD results from combined effects of numerous factors, which have been robustly identified across a variety of research fields, including psychiatry, sociology, and neurobiology. This plurality is embodied in a comprehensive theoretical framework, the biopsychosocial model of addiction, composed of elements whose effects have been well defined individually, but remain poorly characterized and understood in combination. More recently, behavioral epigenetics has emerged as a promising discipline to identify molecular mechanisms that may help explain how life experiences, in particular psychiatric and sociological factors, modulate the regulation of genes, brain function, and emotional regulation. In this context, here we propose a multidisciplinary project that builds on the collaboration of psychiatrists, sociologists and neuro-epigeneticists. The investigators will simultaneously characterize major psychiatric and social factors in a large cohort of individuals with OUD, with the goal of covering the full spectrum of disease severity. By combining deep psychosocial evaluation with the investigation of blood-derived epigenetic biomarkers, they will seek to provide a new and deeper understanding of determinants of OUD severity.

The project builds on 3 main hypotheses:

1. Social and psychiatric factors together contribute to OUD severity;
2. Epigenetic mechanisms, measured in peripheral accessible tissues such as blood, represent biomarkers that may reflect pathophysiological processes resulting, at least in part, from the effects of psychosocial factors;
3. Measures of OUD severity combining both psychosocial factors and epigenetic biomarkers have the potential to improve our ability to describe OUD severity, and better predict its clinical course.

DETAILED DESCRIPTION:
First aim of the study is to systematically characterize OUD severity (DSM-5 criteria) and psychosocial factors in N=350 individuals with OUD, recruited at Safe Injection Sites (SIS), and other addiction-related facilities: French low-risk consumption room (CSAPA), Center for Reception and Accompaniment in Harm Reduction for Drug Users (CAARUD), and pain treatment centers.

Recruitment at SIS will allow to target OUD patients at highest psychosocial risk, who remained mostly out-of-reach of previous studies, and to compare them to stabilized OUD patients, overall covering a wide spectrum of disease course and severity.

Second aim of the study is to examine genome-wide epigenetic regulation (DNA methylation) and gene expression in peripheral blood samples collected from all subjects, at inclusion; then, to leverage systems biology to characterize relationships among these molecular measures and OUD and psychosocial severity;

Third aim of the study is to assess the evolution of OUD and psychosocial severity in the whole cohort, over 2 years, in order to determine how such evolution can be predicted using molecular epigenetic biomarkers defined at inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Male, female, or transgender person, age > 18 years
* French speaking subject, able to understand the objectives and risks of the research
* Informed signed consent form by the curator (subject under curatorship) / guardian (subject under guardianship), if applicable
* Subject who has written "I consent" on the consent form
* Subject using psychoactive substances and who attends a low-risk consumption room (SCMR), or a Center for Care, Accompaniment and Prevention in Addictology (CSAPA), or a Center for Reception and Accompaniment in Harm Reduction for Drug Users (CAARUD)
* Subject who used one or more illegal opioid drugs or one or more medications (with or without a prescription) at least once in the last 3 months (heroin, buprenorphine, morphine sulfate, methadone, morphine derivatives, oxycontin, oxycodone, oxynorm, Subutex® (Sub), Temgesic®, Suboxone®, Orobupre®, Skenan®, Moscontin®, opium, pethidine, codeine, dinacode, neocodion, codeine efferalgan, Lamaline®, tramadol, durogesic patches, fentanyl...)

Exclusion Criteria:

* Inability to give the subject informed information (subject with difficulties in understanding)
* Subject in an emergency or life-threatening situation
* Subject under court protection (upon subject's declaration)
* Subject participating in an investigational drug study (upon subject's declaration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited:
  * in the 2 SIS in Paris (Gaia) and Strasbourg (Ithaque),
  * in French addiction care centers: CAARUD (harm reduction services for drugs users) and CSAPA (primary care outpatient settings for patients with addiction) in Strasbourg, Paris and Lyon
  * in Pain treatment centers in Strasbourg and Lyon.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2029-05-14 (Estimated); Study Completion 2029-05-14 (Estimated)

PRIMARY OUTCOMES:
To systematically characterize OUD severity (DSM -5 criteria ) and psychosocial factors in N=300 individuals with OUD | At inclusion
  Opioid users will be recruitedat Safe Injection Sites (SIS) where we are privileged access, and others addiction related facilities (French CSAPA,CAARUD, and pain treatment centers. Recruitment at SIS will allow the investigators to target OUD patients at highest psychosocial risk, who remained mostly out-of-reach of previous studies, and to compare them to stabilized OUD patients, overall covering a wide spectrum of desease course and severity.

SECONDARY OUTCOMES:
Examine genome -wide epigenic regulation and gene expression in peripheral blood samples collected from all subjects, at inclusion assess the evolution of OUD and psychosocial severity in the cohort, over 2 years. | At inclusion and 24 month after inclusion
  Two secondary outcome will be measured (1) The investigators want to examine genome -wide epigenic regulation (DNA methylation) and gene expression in peripheral blood samples collected from all subjects, at inclusion; then to leverage systems biology to characterize relationships among these molecular measures and OUD and psychosocial severity (2) The investigators want to assess the evolution of OUD and psychosocial severirity in the whole cohort, over 2 years, in order to determine how such evolution can be predicted using molecular epigenic biomarkers defined at inclusion

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service Universitaire d'Addictologie, Hospices Civils de Lyon, Bron
  - Centre d'étude des mouvements sociaux (CEMS) UMR8044/INSERM U1276 - École des Hautes Etudes en Sciences Sociales (EHESS), Paris
  - Service d'Addictologie, Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lalanne L, Lutz PE, Caparros-Roissard A, Ruppert E, Waeckerle G, Scherer C, Oster F, Brand C, Henck S, Soavelo H, Ramousset C, Lebreton M, Audran M, Lazic J, Detrez V, Avril E, Merah I, Chappuy M, Meyer N, Jauffret-Roustide M, Rolland B. Integrative exploration of bio-psycho-social determinants of DSM-5 severity levels of opioid use disorder: the BEBOP cohort study protocol. BMJ Open. 2025 Oct 13;15(10):e093358. doi: 10.1136/bmjopen-2024-093358. PMID 41083308